CLINICAL TRIAL: NCT01166984
Title: Phase 1, Double Blind, Placebo-Controlled, Dose Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Clinical Trial of AB103, A Peptide Antagonist in Healthy Volunteers
Brief Title: AB103 Peptide Antagonist in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atox Bio Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ATB-001
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteer Safety Study
Keywords: sepsis; septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — AB103

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AB103 7.5 µg/kg (Experimental): AB103 7.5 µg/kg administered as a single IV infusion
  Interventions: Drug: AB103
- AB103 37.5 µg/kg (Experimental): AB103 37.5 µg/kg administered as a single IV infusion
  Interventions: Drug: AB103
- AB103 150 µg/kg (Experimental): AB103 150 µg/kg administered as a single IV infusion
  Interventions: Drug: AB103
- AB103 450 µg/kg (Experimental): AB103 450 µg/kg administered as a single IV infusion
  Interventions: Drug: AB103
- Placebo (Placebo Comparator): Normal saline (0.9% sodium chloride) administered as a single IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AB103 — Single intravenous infusion at doses of 7.5 µg/kg, 37.5 µg/kg, 150 µg/kg, or 450 µg/kg administered over approximately 10 minutes
  Arms: AB103 150 µg/kg; AB103 37.5 µg/kg; AB103 450 µg/kg; AB103 7.5 µg/kg
Drug: Placebo — Single intravenous infusion of normal saline (0.9% sodium chloride) administered over approximately 10 minutes
  Arms: Placebo

SUMMARY:
The primary objective of this study is to establish the safety profile and maximum tolerated dose (MTD) of AB103 given as a single intravenous (IV) infusion in healthy volunteers.

DETAILED DESCRIPTION:
After consent and establishing eligibility for the study, each subject received a single IV infusion of escalating doses of AB103 (7.5, 37.5, 150, 450 μg/kg in 5 subjects at each dose) or placebo (n=5). Screening blood chemistry, hematology, coagulation, urinalysis, vital signs, and electrocardiogram (ECG) were used to assure medical fitness to participate in the study. These measures were repeated during and after treatment with AB103 to monitor for adverse events (AEs). ECG and pulse oximetry was monitored continuously starting 15 minutes before the infusion and for 2 hours after each infusion. Vital signs (sitting blood pressure, temperature, heart rate, respiratory rate, and pulse oximetry) and ECG measurements were recorded every 15 minutes for the first two hours starting from the beginning of the infusion and then approximately 24 hours later. Blood chemistry, hematology, coagulation, and urinalysis, were repeated one day and one week after infusions. AEs either observed by the investigator or reported spontaneously by the subjects were recorded at each study visit. Subjects kept a 7-day diary starting on the day of infusion to record any AEs. The primary basis on which escalation was based was dose limiting toxicities (DLTs) defined as the emergence of one or more selected AEs that reached a threshold which justified stopping the trial. After safety monitoring committee review of safety data, progression to the next cohort was to occur as follows:

1. If none of the 5 AB103 subjects in a cohort experienced a non-extreme DLT, escalation to the next dose cohort was to occur.
2. If 1 of 5 subjects receiving AB103 in a cohort experienced a non-extreme DLT, then a total of 8 subjects (6 active: 2 placebo) were to be enrolled in that cohort before escalating to the next dose (escalation will only occur if no additional subjects (2 total) have a non-extreme DLT).
3. If there were 0/6 or 1/6 active subjects with a non-extreme DLT at the highest dose, the highest dose was to be considered the MTD. If there were 2/6 active subjects with a non-extreme DLT in a cohort, then the next lowest dose was to be considered the MTD.
4. If an extreme DLT occurred, the study was to be halted immediately.

Subjects in Cohorts #1 to #3 had a blood sample (40 milliliters, mL) drawn pre-infusion, 24 hours after the infusion (Day 2), and a final sample at the Day 6-8 clinic visit (total of 120 mL) for leukocyte phenotyping by flow cytometry. Subjects in Cohort #4 had a blood sample (40 mL) drawn pre-infusion, 1 hour after the infusion, and a final sample at the Day 6-8 clinic visit (total of 120 mL) for leukocyte phenotyping by flow cytometry.

For the pharmacokinetic (PK) analysis, blood was collected at the mid-point of the infusion and 1, 2, 5, 10, 20, 30, and 60 minutes and approximately 24 hours post-infusion, and plasma was isolated for quantitation of AB103 peptide concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read, understand and sign the Informed Consent form and be willing to participate in all study procedures for the duration of the study.
* Be 18-to-40 years-of-age.
* Have adequate venous access.
* Have a body mass index between 20 and 29 kg/m2.
* Have a history and physical examination that demonstrate no clinically significant contraindication for participating in the study, in the judgment of the admitting physician and/or the site investigator.
* Have vital signs as follows: resting heart rate between 50 and 90 beats per minute (bpm), systolic blood pressure (BP) below 150 mm Hg and diastolic BP below 90 mm Hg.
* Have all blood chemistry, hematology, coagulation, and urinalysis analyte levels within 10% of normal laboratory limits.
* If female, not be pregnant or breast-feeding, nor plan to become pregnant for the duration of the study, have a negative pregnancy test.
* Agree to exercise adequate birth control from the time of the screening procedures to 14 days after the investigational agent administration (both males and females).
* Have an electrocardiogram (ECG) performed that demonstrates normal sinus rhythm, normal conductivity, and no clinically significant arrhythmias.

Exclusion Criteria:

* Be pregnant or lactating.
* Have autoimmune disease or asthma.
* Have been febrile within 3-days of the first infusion.
* Have a history of migraine headaches, as diagnosed by a physician.
* Have any acute or chronic medical illnesses or other condition that, in the opinion of the Investigator, might jeopardize the safety of the patient, or the adequate evaluation of study results.
* Be taking any medications to treat a chronic medical condition.
* Have participated in a research study where they received any experimental products within 30 days prior to study entry.
* Have ongoing drug abuse/dependence (including alcohol) by medical history.
* Have taken, within 14 days of planned dosing, any prescription or non-prescription medication (including ibuprofen, aspirin, of non-steroidal anti-inflammatory drugs) unless the Principal Investigator/Sub-Investigator, in consultation with the Medical Monitor, provides a statement justifying that the medication taken will not impact the results of this study (with rare exceptions taking prescription drugs will be grounds for exclusion).
* Have donated a unit of blood within the preceding 4-week period.
* Have allergy to either sulfa- or penicillin-based drugs.
* Have a history of vagal responses resulting in bradycardia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Cross, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the University of Maryland School of Medicine starting 7 September 2010. The study concluded 10 April 2011.
Pre-assignment Details: One consented and screened subject found to be eligible was not randomized into the study because the target number of subjects had already been achieved.
Groups:
- AB103 7.5 µg/kg: AB103 7.5 µg/kg single IV infusion
- AB103 37.5 µg/kg: AB103 37.5 µg/kg single IV infusion
- AB103 150 µg/kg: AB103 150 µg/kg single IV infusion
- AB103 450 µg/kg: AB103 450 µg/kg single IV infusion
- Placebo: Normal saline (0.9% sodium chloride) single IV infusion
Period: Overall Study
Arm/Group | AB103 7.5 µg/kg | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg | Placebo
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AB103 7.5 µg/kg | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 5 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7) | 29 (6) | 34 (5) | 30 (4) | 30 (8) | 30 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 3 | 1 | 8
  Male | 3 | 4 | 4 | 2 | 4 | 17
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 5 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a subject administered study drug and that does not necessarily have a causal relationship with the study drug. An AE could therefore be any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: 2 weeks
Population: The analysis population consisted of all subjects who received a dose of study drug.
Measure: Number; unit: adverse events
Groups:
- AB103 7.5 µg/kg: Each subject received a single IV infusion of AB103 7.5 µg/kg
- AB103 37.5 µg/kg: Each subject received a single IV infusion of AB103 37.5 µg/kg
- AB103 150 µg/kg: Each subject received a single IV infusion of 150 µg/kg
- AB103 450 µg/kg: Each subject received a single IV infusion of 450 µg/kg
- Placebo: Each subject received a single IV infusion of normal saline (0.9% sodium chloride)
Arm/Group | AB103 7.5 µg/kg | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
adverse events | 7 | 2 | 1 | 9 | 3

2. Primary Outcome: Number of Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is an AE occurring during any study phase and at any dose of the study drug (AB103 or placebo) that fulfills one or more of the following criteria:
  * Results in death
  * Is life-threatening (i.e., the subject was, in the opinion of the Investigator, at immediate risk of death from the event as it occurred)
  * Requires or prolongs hospitalization
  * Results in persistent or significant disability or incapacity (i.e., the event causes a substantial disruption of a person's ability to conduct normal life functions)
  * Is a congenital anomaly or birth defect, or
  * Is an important and significant medical event.
Time Frame: 2 weeks
Population: The analysis population consisted of all subjects receiving a dose of study drug.
Measure: Number; unit: serious adverse events
Groups:
- AB103 7.5 µg/kg: AB103 single IV infusion of 7.5 µg/kg
- AB103 37.5 µg/kg: AB103 single IV infusion of 37.5 µg/kg
- AB103 150 µg/kg: AB103 single IV infusion of 150 µg/kg
- AB103 450 µg/kg: AB103 single IV infusion of 450 µg/kg
Arm/Group | AB103 7.5 µg/kg | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
serious adverse events | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Dose-limiting Toxicities (DLTs)
Description: DLTs were defined as the emergence of one or more selected AEs that reached a threshold that may justify stopping the trial.
Time Frame: 2 weeks
Measure: Number; unit: DLTs
Arm/Group | AB103 7.5 µg/kg | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
DLTs | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC)
Description: Area under the plasma concentration-time curve (AUC) from time zero to infinity following a single dose of study drug, obtained via noncompartmental methods. It is an integrated measure of study drug plasma exposure.
Time Frame: Whole blood was collected pre-dose; at the mid-point of the infusion; at 1, 2, 5, 10, 20, 30, and 60 minutes post-infusion; and at approximately 24 hours post-infusion for the measurement of AB103 plasma concentrations.
Population: AUC could not be determined in the AB103 7.5 µg/kg group and the placebo group because of the number of plasma concentration results that were undetectable.
Measure: Median (Full Range); unit: ng*min/mL
Groups:
- AB103 150 µg/kg: Each subject received a single IV infusion of AB103 150 µg/kg
- AB103 450 µg/kg: Each subject received a single IV infusion of AB103 450 µg/kg
Arm/Group | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg
Number analyzed (Participants) | 5 | 5 | 5
ng*min/mL | 527 [238 to 911] | 2085 [1740 to 2743] | 5831 [4214 to 9441]

5. Secondary Outcome: Cmax
Description: Maximum plasma concentration
Time Frame: as for outcome 4
Population: Cmax is not available (applicable) to placebo patients (no detectable plasma concentrations).
Measure: Median (Full Range); unit: ng/mL
Arm/Group | AB103 7.5 µg/kg | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5
ng/mL | 10.63 [7.35 to 11.97] | 52.67 [19.99 to 104.35] | 190.90 [160.77 to 295.21] | 611.19 [455.36 to 1031.71]

6. Secondary Outcome: Apparent Terminal Plasma Half-life (T1/2)
Description: Apparent terminal plasma half-life (T1/2) is the amount of time for plasma concentrations to decline by 50%.
Time Frame: as for outcome 4
Population: This outcome measure could not be determined in the 7.5 µg/kg dose group because of the frequency of undetectable plasma concentrations. It was not determined for placebo subjects (undetectable plasma concentrations).
Measure: Median (Full Range); unit: hours (h)
Arm/Group | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg
Number analyzed (Participants) | 5 | 5 | 5
hours (h) | 1.42 [0.78 to 1.83] | 1.36 [0.77 to 1.48] | 1.28 [1.16 to 1.67]

7. Secondary Outcome: Clearance (CL)
Description: Clearance (CL) is the volume of plasma completely cleared of drug per unit of time.
Time Frame: as for outcome 4
Population: Clearance was not determined in the 7.5 µg/kg dose group because of the frequency of undetectable AB103 plasma concentrations. Clearance was not determined in the placebo group (undetectable plasma concentrations).
Measure: Median (Full Range); unit: mL/min/kg
Arm/Group | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg
Number analyzed (Participants) | 5 | 5 | 5
mL/min/kg | 71 [41 to 158] | 72 [55 to 86] | 77 [48 to 107]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | AB103 7.5 µg/kg | AB103 37.5 µg/kg | AB103 150 µg/kg | AB103 450 µg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5 | 1/5 | 2/5 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AB103 7.5 µg/kg (N=5) | AB103 37.5 µg/kg (N=5) | AB103 150 µg/kg (N=5) | AB103 450 µg/kg (N=5) | Placebo (N=5)
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pruritis genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No